CLINICAL TRIAL: NCT00704119
Title: CT 5002 An Open-label, Non-randomized, Monocentric Phase I Study Evaluating the Pharmacokinetic Profile of RhuDex® Using a Tablet Formulation
Brief Title: Study Evaluating the Pharmacokinetic Profile of RhuDex® in a Tablet Formulation
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Following an SAE, study was put on hold. After performing preclinical follow-up studies, volunteers were no longer available for continuation.
Sponsor: MediGene (Industry)
Responsible Party: Prof. HodaTawfik, Clinical Project Manager, MediGene AG
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: CT 5002
Record Dates: First submitted 2008-06-23; First posted 2008-06-24 (Estimated); Last update posted 2010-03-24 (Estimated); Status verified 2010-03

CONDITIONS: Pharmacokinetics
Keywords: Rhudex; pharmacokinetic study

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: RhuDex® — * Treatment A.1: 31.65 mg RhuDex® once N=12
  * Treatment A.2: 63.33 mg RhuDex® once N=12
  * Treatment A.3: 126.63 mg RhuDex® once N=12
  * Treatment A.4: 253.26 mg RhuDex® once N=12
  * Treatment B.1: 31.65 mg RhuDex® once N=12
  * Treatment B.2: selected dose of RhuDex® once N=12
  * Treatment C: selected dose of RhuDex® once N=12
  * Treatment D: selected dose of RhuDex® twice daily for 6 days N=12
  Other Names: AV1142742

SUMMARY:
RhuDex® (code number AV1142742) is a novel, orally bioavailable, low molecular weight modulator of co-stimulation of T lymphocytes. RhuDex® binds to the protein CD80 (also known as B7-1) on the surface of antigen-presenting cells and inhibits its interaction with CD28 (but not with CTLA-4) presented by CD4+ T lymphocytes.

RhuDex® is being developed for the treatment of rheumatoid arthritis. To improve oral bioavailability, the study drug has to be co-administered with an alkaline buffer that increases gastric pH values. In previous in vitro and phase I studies, meglumine has been identified as the most effective buffer. Study CT 5002 is designed to evaluate the bioavailability of four increasing doses of RhuDex®, combined with a fixed amount of meglumine using a tablet formulation, under fed and fasted conditions as well as with co-administration of the proton pump inhibitor pantoprazole. Furthermore, dose/plasma concentration proportionality for single dosing and accumulation effects for repeat dosing of RhuDex® will be evaluated.

DETAILED DESCRIPTION:
This is an open-label, non-randomized, monocentric Phase I study to evaluate the pharmacokinetic profile of single-dosed and repeat-dosed RhuDex® using a tablet formulation as well as to assess the effect of food and the effect with co-administration of a proton pump inhibitor on the bioavailability of RhuDex®.

12 healthy male subjects will receive study medication in 8 different treatment periods in 4 subsequent steps A, B, C and D.

Within steps A and B, the subjects will receive different treatments (4 in A and 2 in B), sequentially. There will be a wash-out period of at least 4 days between each of the 8 different treatments/treatment periods of steps A, B, C and D.

In Step A, each subject will receive increasing doses of RhuDex® in 4 subsequent treatments. In Step B, each subject will receive 2 different doses of RhuDex® preceded by pantoprazole intake, in 2 subsequent treatments, and in Step C the RhuDex® dosing will be preceded by a standardized high-fat, high-calorie meal. In Step D, RhuDex® will be administered twice daily for 7 days.

For assessing the pharmacokinetic profile of RhuDex® in steps A, B and C, blood samples will be collected prior to and at different intervals after RhuDex® administration. In step D, blood samples will be collected on Days 1, 2, 4 and 7. Cmin, Cmax, tmax, t½ term, CL/F, AUC(0-t), and AUC(0-∞) of RhuDex® will be analyzed.

Safety will be evaluated by regular observation and documentation of AEs, vital signs, physical examination, ECG, and laboratory parameters.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male subjects between 18 and 60 years at the time of enrolment
2. Subjects who are sexually active must use adequate contraception for the duration of the study from screening until 12 weeks after the last dose.
3. BMI between 18.5 and 29.9 kg/m²
4. Written informed consent
5. Ability to comply with the requirements of the study

Exclusion Criteria:

1. Acute infection at time of enrolment
2. History of chronic inflammation, chronic infection, other chronic disease, autoimmune disorders (e.g. diabetes mellitus) or cancer
3. Clinically significant abnormal ECG
4. Clinically significant abnormal laboratory values (especially in terms of liver or renal insufficiency)
5. Clinically significant physical findings
6. Major surgery within the last 4 weeks prior to enrolment
7. Organ allograft recipient
8. Concomitant or planned treatment which would interfere with study results
9. Any systemic medical treatment, including over the counter products and dietary supplements such as iodine, fluoride or vitamins, within one week before and during the study course
10. Known allergy against any ingredient of the study medication, meglumine, pantoprazole or bovine milk
11. Participation in an investigational trial within 12 weeks prior to enrolment
12. Systemic intake of immunosuppressive or immunomodulatory medication or vaccination within 30 days prior to enrolment and for the whole study duration
13. Blood loss exceeding 450 mL (including blood donations) within 12 weeks prior to enrolment into the study.
14. Medical history of alcohol or drug abuse within the last 2 years or alcohol consumption greater than 21 units per week.
15. A positive alcohol breath test
16. A positive urine drug screen
17. Smokers who smoke > 5 cigarettes or 5 cigars per day
18. Presence of hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCV Ab) or HIV-1 or HIV-2 antibodies at screening
19. Subject whose partner is pregnant or lactating

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2008-05; Primary Completion 2008-07 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
To assess the relationship between the dose of RhuDex® administered and the plasma concentrations achieved following single and repeated doses under fed and/or fasted conditions and with/without administration of pantoprazole | 24 -96h pharmakokinetic laboratory values

SECONDARY OUTCOMES:
To gain further safety and tolerability data of RhuDex® | during treatment phase and 28 days afterwards

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Mair, MBChB, DROCG,DCPSA, Principal Investigator — Syneos Health
Locations (1):
- Charles River Clinical Services Edinburgh Ltd, Edinburgh, Scotland, United Kingdom